CLINICAL TRIAL: NCT05292235
Title: A Prospective Assessment of the Perioperative Parameter and Treatment Outcomes of Surgical Treatment for Benign Prostate Hyperplasia in Hong Kong
Brief Title: Perioperative Parameter and Treatment Outcomes of Surgical Treatment for Benign Prostate Hyperplasia in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2022.049
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective data registry to assess the treatment outcomes and complications of different treatment approaches in our hospital clusters.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a very common disease affecting men. Patients with BPH may present with voiding symptoms including hesitancy, intermittence, slow stream and sensation of incomplete emptying, and storage symptoms including urinary frequency, urgency and nocturia. Patients may also suffer from complications including urinary retention, recurrent urinary tract infection, bladder stone formation and obstructive uropathy. For patients who have lower urinary tract symptoms refractory to medications, or those who suffer from complications of BPH, transurethral prostatectomy should be considered.

Surgical intervention options have evolved from electrosurgical resection to the use of lasers for enucleation and ablation [1]. Aquablation and Rezum system are new minimally invasive surgical technology for BPH management. [2,3,4]. Different treatment approaches will result in different treatment successful rate and also potential adverse effects to patients.

However, large-scale studies investigating the different modalities of surgical treatment of BPH are lacking. Therefore, a prospective data registry is created to assess the perioperative surgical outcomes for different surgical treatment of BPH.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the age of 18 or above

Exclusion Criteria:

* Patient is unable to give consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with BPH and planned for surgery (including all type of endoscopic procedures) in the hospitals will be identified and then enrolled to the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2032-04-30 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) questionnaire total Score | Baseline, 3 months after surgical treatment for BPH
  Change in total scores in International Prostate Symptom Score (ranges from 0 to 35) questionnaires
Voiding function in uroflowmetry | Baseline, 3 months after after surgical treatment for BPH
  Change in urodynamic function assessed by Uroflowmetry

SECONDARY OUTCOMES:
Complication after surgical treatment | Post operation 30 days after surgical treatment for BPH
  The 30-day complications will be graded according to the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - North District Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahokehr A, Gilling PJ. Landmarks in BPH--from aetiology to medical and surgical management. Nat Rev Urol. 2014 Feb;11(2):118-22. doi: 10.1038/nrurol.2013.318. Epub 2014 Jan 21. PMID 24445912
- [Background] Magistro G, Chapple CR, Elhilali M, Gilling P, McVary KT, Roehrborn CG, Stief CG, Woo HH, Gratzke C. Emerging Minimally Invasive Treatment Options for Male Lower Urinary Tract Symptoms. Eur Urol. 2017 Dec;72(6):986-997. doi: 10.1016/j.eururo.2017.07.005. Epub 2017 Jul 19. PMID 28734706
- [Background] Faber K, de Abreu AL, Ramos P, Aljuri N, Mantri S, Gill I, Ukimura O, Desai M. Image-guided robot-assisted prostate ablation using water jet-hydrodissection: initial study of a novel technology for benign prostatic hyperplasia. J Endourol. 2015 Jan;29(1):63-9. doi: 10.1089/end.2014.0304. PMID 25000418
- [Background] Dixon CM, Rijo Cedano E, Mynderse LA, Larson TR. Transurethral convective water vapor as a treatment for lower urinary tract symptomatology due to benign prostatic hyperplasia using the Rezum((R)) system: evaluation of acute ablative capabilities in the human prostate. Res Rep Urol. 2015 Jan 30;7:13-8. doi: 10.2147/RRU.S74040. eCollection 2015. PMID 25674555